CLINICAL TRIAL: NCT06856239
Title: Comparison of Flexural Strength and Flexural Modulus of Conventional and Graphene-Reinforced Polymethyl Methacrylate
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Altamash Institute of Dental Medicine (Other)
Responsible Party: Principal Investigator, Wajiha Zia, Prinicipal investigator, Altamash Institute of Dental Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AltamashWZ
Record Dates: First submitted 2025-02-10; First posted 2025-03-04 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Dentures; Denture,Complete
MeSH Terms: interventions — Graphite

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PMMA(polymethyl methacrylate) (No Intervention): Polymethyl methacrylate (PMMA), which was invented by Dr. Walter Wright1 in 1937, and is now one of the most widely used denture base materials. Polymethyl methacrylate (PMMA) has gained popularity due to its low cost, adequate mechanical strength, acceptable aesthetics, good dimensional stability, and biocompatibility. However, it has low flexural strength, fatigue fracture, and impact strength which can lead to fracture of the prosthesis.
- G-PMMA( Graphene-polymethyl methacrylate) (Experimental): Graphene was first invented by Novoselov et al,16 Graphene is a two dimensional (2D), monolayer sp2 hybridized carbon atoms and recognized as the thinnest material in the universe. Comparing it to other traditional nanofillers, its large surface area, tensile strength, flexibility, strong thermal and electrical conductivity, and low coefficient of thermal expansion give it a better result.17 Recent studies have discovered that graphene and its derivatives, which include graphene oxide and reduced graphene oxide, have better outcomes as compared to conventional materials
  Interventions: Other: Graphene

INTERVENTIONS:
Other: Graphene — The study follows an in-vitro experimental design with 76 specimens divided into two groups (conventional PMMA and G-PMMA). These samples will be further divided into two group, the one which undergo thermocycling (simulating oral temperature changes) and the other which don't undergo thermocycling. Flexural strength and modulus will be tested on all these by using a three-point bending test.
  Arms: G-PMMA( Graphene-polymethyl methacrylate)

SUMMARY:
Study Title: Comparison of Flexural Strength and Modulus of Conventional and Graphene-Reinforced PMMA

Introduction:

This in-vitro experimental study aims to compare the flexural strength and flexural modulus of conventional polymethyl methacrylate (PMMA) and graphene-reinforced PMMA (G-PMMA) used in denture bases. PMMA is widely used for dentures due to its affordability, aesthetics, and biocompatibility but has limitations such as low flexural strength and susceptibility to fracture. Graphene, a strong and flexible nanomaterial, has demonstrated potential in enhancing PMMA's mechanical properties.

OBJECTIVE:

To compare the flexural strength and flexural modulus of conventional and graphene reinforced polymethyl methacrylate

HYPOTHESIS:

Null Hypothesis:

There is no difference in flexural strength and flexural modulus of graphene reinforced PMMA and conventional PMMA.

Alternative Hypothesis:

There is a difference in flexural strength and flexural modulus of graphene-reinforced PMMA and conventional PMMA.

Methodology:

* Study Design: In-vitro experimental trial
* Study SETTING:

  * The study will be carried out at Altamash Institute of Dental Medicine in the department of prosthodontic, Karachi Pakistan.
  * The graphene (Miraculum Graphene Private Limited,Gujrat, Ahmedabad,India) will be reduced at Karachi University's Food Science Department.
  * For the formation of mold, the digital metal bar (CoCr, Eplus3D, Hangzhou China) will be fabricated by Selective laser melting (SLM) (Audental Shanghai, East-central China) at Chughtai Lab in Peshawar, Pakistan.
  * The acrylic (Mr. Teeth, Royale Elite, Surrey,United Kingdom) samples will be cured by short curing cycling in the prosthodontic department at Bahria dental University, Karachi.
  * The thermocycling (thermocycler, San Francisco, USA) and universal testing for flexural strength and modulus of acrylic samples will be performed at the research laboratory of Dow University of health sciences.
* Sample Size: The projected sample size for this study is 76 specimen, 38 samples per group by comparing two means in open epi software19 (version 3).The calculation was based on the result of Kaan Yerliyurt 11 study, considering the mean value of 68.16 MPa and standard deviation (SD) of 5.79 MPa for the experimental group and the mean value of 72.6 MPa and standard deviation (SD) of 7.84 MPa for the control group of flexural strength. The analysis accounts for multiple time intervals, and the significance level (α) is set at 0.05, with a power of 80%, confidence interval (CI) of 95%, a margin of error (ME) of 5%.

  76 specimens (38 for conventional PMMA, 38 for G-PMMA)
* Subgroups: Each group will have thermocycled and non-thermocycled samples to assess durability.

SAMPLING TECHNIQUE:

Stratified sampling followed by systematic division.

* Methodology:
* Thermocycling: 2000 cycles (5°C-55°C) simulating oral temperature variations

Data Collection:

A metal bar mold (65 mm × 10 mm × 3 mm) will be designed using Exocad CAD software and 3D-printed from CoCr material using Selective Laser Melting (SLM). After fabrication, the bar will be used to create a silicone mold, which will then be invested in dental plaster to prepare the final mold for specimen curing. Graphene oxide (GO) will be chemically reduced, purified, dried, and mixed into PMMA powder. The acrylic resin will then be packed into the mold and processed via short curing cycle (74°C for 2 hours, 100°C for 1 hour). Then all the specimen will be prepared, thermocycle and ready for flexural strength and flexural modulus.

- Data Analysis: The data will be evaluated using the statistical package for social sciences (SPSS version 29, IBM, Chicago, Illinois United States). Descriptive statistics will be evaluated by mean, standard deviation, median, interquartile range of flexural strength, flexural modulus for PMMA, and GPMMA. Shapiro-Wilk test will be used to check the normality of the data distribution. For interferential statistics, Kruskal Wallis or ANOVA will be used with factors of loading force (N) and deflection (Y) between G-PMMA and conventional PMMA. Post-hoc analysis will be performed by Bonferroni or Tukey's test. In order to assess the effect of the external environment, the cofounding variable in this study will be thermocycling, which will influence the flexural strength and flexural modulus of PMMA and graphene-reinforced PMMA samples. A Chi-square or independent t-test will be used to analyze the impact of the cofounding variable, thermocycling, on flexural strength and modulus. The level of significance will be set at p < 0.05.

Rationale:

This study aims to determine whether graphene reinforcement improves the mechanical properties of PMMA, potentially leading to stronger and more fracture-resistant dentures. The findings could contribute to the development of more durable denture base materials with enhanced longevity and performance.

ELIGIBILITY:
Inclusion Criteria:

* INCLUSION CRITERIA:

  * Samples that are dimensionally accurate in accordance to ISO Standard 178.21
  * Sample that are free from surface porosities like gaseous, granular or contraction porosities.
  * Samples have uniform color and surface texture indicating proper curing.
  * Samples free from crazing defects and warpage.
  * Samples with no signs of distortion after thermocycling.
  * Samples with homogeneously distributed graphene by visual inspection of samples.

Exclusion Criteria:

* • Samples with incorrect mixing ratio of base to catalyst.

  * Samples in which the metal bar is partially exposed.
  * Samples that are not fully embedded in plaster.
  * Samples showing sign of contamination from foreign body during packing process.
  * Samples with improper mixing of plaster shows a sign of cracks and voids surrounding the samples.
  * Samples in which the flask will not properly sealed during flasking.
  * Samples fractured due to thermocycling.
  * Samples fractured during handling or transportation before testing.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-12-25 (Estimated); Study Completion 2026-01-25 (Estimated)

PRIMARY OUTCOMES:
Flexural strength and Flexural modulus | 1 year
  Outcome Measure 1: Flexural Strength (MPa) The flexural strength of the specimens will be measured using a three-point bending test on a universal testing machine (Testometric testing machine, model VB50-300, Rochdale, Greater Manchester, United Kingdom).
  A load of 0N at a crosshead speed of 2 mm/min will be applied. The force will be increased until the specimens fracture. The maximum force (N) applied before fracture will be recorded to calculate the flexural strength (MPa).
  Outcome Measure 2: Flexural Modulus (MPa) The flexural modulus of the specimens will be tested using a universal testing machine (Testometric testing machine, model VB50-300, Rochdale, Greater Manchester, United Kingdom).
  A constant load of 0N at a crosshead speed of 2 mm/min will be applied. The load (N) and deflection (Y) will be recorded using WinTest software. The initial slope of the load-deflection curve (elastic region) will be used to determine flexural modulus (MPa).

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Naseer Ahmed, Bds,Fcps,PhD, Study Director — Altamash Institute of Dental Medicine
Locations (2):
- Pakistan (2):
  - Altamash institute of dental medicine, Karachi, Sindh
  - Altamash institute of dental medicine, Karachi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Di Carlo S, De Angelis F, Brauner E, Pranno N, Tassi G, Senatore M, Bossu M. Flexural strength and elastic modulus evaluation of structures made by conventional PMMA and PMMA reinforced with graphene. Eur Rev Med Pharmacol Sci. 2020 May;24(10):5201-5208. doi: 10.26355/eurrev_202005_21301. PMID 32495852